CLINICAL TRIAL: NCT00200486
Title: Molecular and Genomic Profiling of Head and Neck Tumors to Explore Biomarkers Associated With Prognosis and Response to Therapy
Brief Title: Molecular and Genomic Profiling of Head and Neck Tumors
Status: Recruiting | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 02-05-127E; NIH-R21-CA104402; 6R21DE023941-03 (NIH); 3P50DE019032-14S2 (NIH); 3U54CA274321-02S1 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Neoplasms
Keywords: genetic microarray; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Tumor specimens along with normal mucosa obtained at the time of surgery for biopsy or resection of primary or recurrent tumors of the head and neck
  2. blood, urine and sputum from patients participating in the tumor collection described above
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to study the genetic profile of head and neck tumors and their relationship to treatment response and outcome

DETAILED DESCRIPTION:
Previous research by our group using genetic microarray analysis of HNSCC and normal keratinocytes has identified two distinct groups of genetic expression based on clustering patterns of a subgroup of genes. Clinical data was summarized for each group and overall, patient segregation by gene expression profiling was a better predictor of outcome than clinicopathological variables. Further analysis identified 375 genes that discriminate between the genotypic subtypes of HNSCC. Overall, our preliminary data has shown that the pattern of global gene expression in a HNSCC specimen can be used as a predictor of prognosis. We isolated subsets of genes showing the greatest patterns of divergence in gene expression. We have also identified 366 over-expressed and 246 underexpressed genes when comparing primary tumor to normal surgical margins and have identified a similar number of genes whose expression has changed when comparing primary tumor to lymph node metastasis. Combining these data sets we have identified genes which consistently increase or decrease expression during progression from normal tissue to primary tumor, and subsequently to metastatic node. We have selected several candidate genes for subsequent analysis using HNSCC tissue arrays. Through DNA microarray analysis and other techniques for looking at genetic and molecular characteristics, a more detailed knowledge of the malignant transformation process, and alterations with therapy, in these patients may be obtained. This study will seek to perform comprehensive molecular and genetic profiling to improve biomarker development in HNSCC and correlate this data with patient clinical data. Ultimately it is hoped that tumor specific genetic abnormalities may be identified which could provide targets for treatment strategies such as gene therapy, immunotherapy, or other interventions.

Study Objectives:

To evaluate gene expression patterns in human head and neck squamous cell carcinoma and correlate this with treatment response, both surgical and non-surgical.

To identify a series of diagnostic markers in blood, urine and/or sputum for head and neck squamous cell carcinoma and study the mechanism of action of these proteins.

ELIGIBILITY:
Inclusion Criteria:

* actual or suspected malignant or non-malignant tumors of the head and neck
* planned biopsy and/or resection, or availability of paraffin embedded or stored frozen tumor tissue for non-genetic analysis

Exclusion Criteria:

* insufficient tissue available for both standard diagnostic evaluation and study specimen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with tumors of the head and neck who ar ehaving diagnostic biopsy or surgical resection of primary lesions or recurrences
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2002-10-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
correlation of treatment response and prognosis (time to recurrence and survival) with genetic expression profile | 5 years

SECONDARY OUTCOMES:
identify a series of diagnostic markers for head and neck tumors and study the mechanism of action of these proteins | variable

CONTACTS AND LOCATIONS:
Overall Officials: Richard V Smith, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Stelby Augustine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stone A, Liu J, Lin J, Schiff BA, Ow TJ, Mehta V, Smith RV. Value of Adherence to Posttreatment Follow-Up Guidelines for Head and Neck Squamous Cell Carcinoma. Laryngoscope. 2024 Feb;134(2):708-716. doi: 10.1002/lary.30909. Epub 2023 Jul 26. PMID 37493178
- [Result] Shrivastava N, Chavez CG, Li D, Mehta V, Thomas C, Fulcher CD, Kawachi N, Bottalico DM, Prystowsky MB, Basu I, Guha C, Ow TJ. CDK4/6 Inhibition Induces Senescence and Enhances Radiation Response by Disabling DNA Damage Repair in Oral Cavity Squamous Cell Carcinoma. Cancers (Basel). 2023 Mar 28;15(7):2005. doi: 10.3390/cancers15072005. PMID 37046664
- [Result] Li D, Thomas C, Shrivastava N, Gersten A, Gadsden N, Schlecht N, Kawachi N, Schiff BA, Smith RV, Rosenblatt G, Augustine S, Gavathiotis E, Burk R, Prystowsky MB, Guha C, Mehta V, Ow TJ. Establishment of a diverse head and neck squamous cancer cell bank using conditional reprogramming culture methods. J Med Virol. 2023 Feb;95(2):e28388. doi: 10.1002/jmv.28388. PMID 36477880